CLINICAL TRIAL: NCT02111876
Title: Systematic Follow-up of Patients Surviving an Episode of Acute Hypercapnic Respiratory Failure in the ICU
Status: Completed | Type: Observational
Sponsor: Ligue Pulmonaire Genevoise (Other)
Collaborators: University Hospital, Geneva (Other)
Responsible Party: Sponsor
Other Study IDs: CE 11-238; LIgue Pulmonaire Genevoise (Other Grant/Funding Number: Ligue Pulmonaire Genevoise)
Record Dates: First submitted 2014-03-10; First posted 2014-04-11 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2014-04

CONDITIONS: Acute Hypercapnic Respiratory Failure
Keywords: ICU, COPD, OHS, OSA, heart failure
MeSH Terms: conditions — Respiratory Insufficiency; Pulmonary Disease, Chronic Obstructive; Sleep Apnea, Obstructive; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- AHRF follow-up

SUMMARY:
There is currently no good description of patients surviving an episode of acute hypercapnic respiratory failure in the ICU. For instance, the prevalence of OSA and sleep hypoventilation in a stable clinical condition is not known in this population.

This prospective cohort describes the clinical profile, predictors of readmission (followed over a year), and the prevalence of sleep-related breathing disorders (polysomnography in a stable clinical condition 3 months after ICU discharge) in patients treated for an episode of acute hypercapnic respiratory failure in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years Informed consent surviving an episode of acute hypercapnic respiratory failure

Exclusion Criteria:

* iatrogenic hypercpania pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients surviving an episode of acute hypercapnic respiratory failure in the ICU
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Sleep apnea syndrome | at 2 month after ICU discharge
  Apnea-Hypopnea Index defined by polysomnography
Sleep Hypoventilation | at 2 month after ICU discharge
  defined by AASM 2012 criteria with transcutaneous PtCO2 monitoring

SECONDARY OUTCOMES:
Lung physiology ( obstructive or restrictive lung disease) | at week 2 after ICU discharge
  FEV1, VC, TLC, DLCO
Inspiratory Muscle Strength | at week 2 after ICU discharge
  Sniff nasal maximal inspiratory pressure, Mouth inspiratory pressure
Cardiac function | at week 2 after ICU discharge
  Systolic and diastolic cardiac function, pulmonary hypertension
Hospital and ICU readmission rate | 1 year follow-up after ICu discharge

CONTACTS AND LOCATIONS:
Overall Officials: Adler E Adler, M.D., Principal Investigator — HUG
Locations (1):
- Hôpitaux Universitaires de Genpve, Geneva, Switzerland

REFERENCES:
- [Derived] Karege G, Zekry D, Allali G, Adler D, Marti C. Gait speed is associated with death or readmission among patients surviving acute hypercapnic respiratory failure. BMJ Open Respir Res. 2020 Jun;7(1):e000542. doi: 10.1136/bmjresp-2019-000542. PMID 32561512
- [Derived] Adler D, Pepin JL, Dupuis-Lozeron E, Espa-Cervena K, Merlet-Violet R, Muller H, Janssens JP, Brochard L. Comorbidities and Subgroups of Patients Surviving Severe Acute Hypercapnic Respiratory Failure in the Intensive Care Unit. Am J Respir Crit Care Med. 2017 Jul 15;196(2):200-207. doi: 10.1164/rccm.201608-1666OC. PMID 27973930